CLINICAL TRIAL: NCT03790917
Title: Assessment of Adherence to New Oral anTicoagulants in Atrial Fibrillation patiEnts Within the Outpatient registrY Profile. Prospective Observational Study. ANTEY Study
Brief Title: Assessment of Adherence to New Oral anTicoagulants in Atrial Fibrillation patiEnts Within the Outpatient registrY
Acronym: ANTEY
Status: Completed | Type: Observational
Sponsor: National Research Center for Preventive Medicine (Other Government)
Responsible Party: Sponsor
Organization: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Other Study IDs: ANTEY
Record Dates: First submitted 2018-12-28; First posted 2019-01-02 (Actual); Results first posted 2020-06-09 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-05

CONDITIONS: Atrial Fibrillation
Keywords: adherence; new oral anticoagulants (NOACs); AF
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A prospective non-interventional single-centre study aimed to evaluate actual adherence of AF patients using the validated adherence Scale.

Primary Study Objective(s) Primary study objective The aim of the present study is to assess adherence to therapy and factors associated with adherence in patients with CV disease complicated by non-valvular atrial fibrillation requiring OAC treatment within the outpatient registry PROFILE (prospective, observational study).

1. Data collection in patients with non-valvular atrial fibrillation requiring OAC treatment included in the registry
2. Evaluation of actual patient adherence to OACs

Secondary Study Objective(s)

1. Evaluation of potential patient adherence to OACs
2. Determination of the most significant factors associated with adherence to OACs in patients with non-valvular AF
3. Validation of new original 5-item Questionnaire
4. Evaluation of doctor's adherence to OAC prescription according to Guidelines (ESC). Management of atrial fibrillation,2016)

DETAILED DESCRIPTION:
AF patients from ongoing PROFILE registry will be invited to visit the scientific center.

2 visits with a 6-month interval are expected for each patient as part of routine clinical practice and phone contact is scheduled for each patient 1 year from the first visit to the scientific center (follow-up period).

ELIGIBILITY:
Inclusion Criteria:

* Men and women above 18 years of age who were included in the PROFILE registry by the start of the observational study
* Presence of written informed consent to participate in the study, fill in the study questionnaires and have personal data analyzed
* Presence of any form of non-valvular atrial fibrillation with CHA2DS2-VASc score of ≥1 or patients with CHA2DS2-VASc score = 0, who are already taking OAK

Exclusion Criteria:

* Patients with high bleeding risk, including patients with:

  * Congenital or acquired bleeding disorders
  * Uncontrolled resistant hypertension
  * Exacerbation of gastric and duodenal ulcer
  * Vascular retinopathy
  * Recent history of intracranial or intracerebral hemorrhage
  * Pathology of the brain and spinal cord vessels
  * Recent history of brain, spinal cord or eye surgery
  * History of bronchiectasis or pulmonary hemorrhage
  * A CHA2DS2-VASc score of 0 (OACs are not indicated)
  * Pregnancy, lactation
  * Planned surgery
  * Known hypersensitivity to ingredients of medications used in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary patients with non-valvular atrial fibrillation included in the outpatient registry PROFILE during the period 01.01.2011-31.08.2015.
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2018-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Martsevich, MD,PhD, Principal Investigator — National Research Center of Preventive Medicine
Locations (1):
- National Research Center for Preventive Medicine, Moscow, Russia

RESULTS

PARTICIPANT FLOW:
Groups:
- ANTEY: Patients with AF from the "PROFILE" registry were included. The study consisted of two visits half a year apart (V0, V1) and a phone contact (PC) one year after V0. During V0 all patients were recommended to start therapy with one of the NOACs. Adherence to therapy was assessed during all visits with the use of the original questionnaire - National society of evidence-based pharmacotherapy (NSEPh) adherence scale and direct doctors' questioning.
Period: Overall Study
Arm/Group | ANTEY
Started | 201
Completed | 200
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | ANTEY
Number analyzed (Participants) | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.1 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83
  Male | 118
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 201
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 201
NOAC recommended to patients by doctors during V0 [Count of Participants; unit: Participants]
  rivaroxaban | 111
  dabigatran | 47
  apixaban | 43

OUTCOME MEASURES:

1. Primary Outcome: Proportions of Adherent, Partially Adherent, Partially Non-adherent and Completely Non-adherent Patients (NSEPh During V1)
Description: The study consisted of two visits half a year apart (V0, V1) and a phone contact (PC) one year after V0. During V0 all patients were recommended to start therapy with one of the NOACs.
  Adherence to therapy was assessed during V1 with the use of the original questionnaire - National society of evidence-based pharmacotherapy (NSEPh) adherence scale.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- ANTEY: Patients with AF from the "PROFILE" registry were included. The study consisted of two visits half a year apart (V0, V1) and a phone contact (PC) one year after V0. During V0 all patients were recommended to start therapy with one of the NOACs. Adherence to therapy was assessed during all visits with the use of the original questionnaire - National society of evidence-based pharmacotherapy (NSEPh) adherence scale, 8-item Morisky Medical Adherence Scale (MMAS-8) and direct doctors' questioning.
Arm/Group | ANTEY
Number analyzed (Participants) | 200
Participants
  completely adherent | 155
  partially adherent | 5
  partially non-adherent | 7
  completely non-adherent | 33

2. Primary Outcome: Proportions of Adherent, Partially Adherent, Partially Non-adherent and Completely Non-adherent Patients (NSEPh During Phone Contact)
Description: The study consisted of two visits half a year apart (V0, V1) and a phone contact (PC) one year after V0. During V0 all patients were recommended to start therapy with one of the NOACs.
  Adherence to therapy was assessed during phone contact with the use of the original questionnaire - National society of evidence-based pharmacotherapy (NSEPh) adherence scale.
  Out of 201 participants of the study 4 patients died and 197 patients completed the study.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | ANTEY
Number analyzed (Participants) | 197
Participants
  completely adherent | 158
  partially adherent | 6
  partially non-adherent | 18
  completely non-adherent | 15

3. Secondary Outcome: Proportion of Potentially Adherent Patients
Description: Specifically designed 5-item questionnaire was used for assessment of potential adherence to OACs. According to results patients were divided into groups: completely adherent, partially adherent, completely non-adherent to OACs.
Time Frame: Total - 1 year (two timepoints - 6 months (V1) and 1 year (PC)
Measure: Count of Participants; unit: Participants
Arm/Group | ANTEY
Number analyzed (Participants) | 201
Participants
  completely adherent | 161
  partially adherent | 28
  completely non-adherent | 12

4. Secondary Outcome: Proportion of OACs Prescribed by Doctors According to Guidelines
Description: Prescription of OACs according to guidelines was considered "positive" if it matched the key points of 2016 ESC Guidelines for the management of atrial fibrillation.
  1. Oral anticoagulation therapy to prevent thromboembolism is recommended for all male AF patients with a CHA2DS2-VASc score of 2 or more.
  2. Oral anticoagulation therapy to prevent thromboembolism is recommended in all female AF patients with a CHA2DS2-VASc score of 3 or more.
  3. Antiplatelet monotherapy is not recommended for stroke prevention in AF patients, regardless of stroke risk.
  4. NOACs (apixaban, dabigatran, edoxaban, and rivaroxaban) are not recommended in patients with mechanical heart valves (Level of evidence B) or moderate-to-severe mitral stenosis (Level of evidence C).
  5. In male or female AF patients without additional stroke risk factors, anticoagulant or antiplatelet therapy is not recommended for stroke prevention.
Time Frame: Total - 1 year (two timepoints - 6 months (V1) and 1 year (PC)
Measure: Count of Participants; unit: Participants
Arm/Group | ANTEY
Number analyzed (Participants) | 201
Participants
  OACs were recommended by doctors | 171
  OACs were not recommended by doctors | 30

5. Secondary Outcome: The Main Reasons for Refusing to Start NOAC Therapy
Description: The study consisted of two visits half a year apart (V0, V1) and a phone contact (PC) one year after V0. During V0 all patients were recommended to start therapy with one of the NOACs. Patients refusing to start NOAC treatmet were asked about the reasons to refuse NOAC treatment.
Time Frame: Total - 1 year (two timepoints - 6 months (V1) and 1 year (PC)
Measure: Count of Participants; unit: Participants
Arm/Group | ANTEY
Number analyzed (Participants) | 33
Participants
  high price of NOAC | 14
  fear of adverse events | 6
  doubts about the correctness of prescribtion | 5
  adherence to Warfarin | 2
  adherence to another NOAC | 2
  difficult regimen for all drugs | 2
  lack of NOAC in the preferential drug list | 2

6. Secondary Outcome: Reasons for Stopping Oral Anticoagulants (Data From Visit 1)
Description: The study consisted of two visits half a year apart (V0, V1) and phone contact (PC) one year after V0. During V0 all patients were recommended to start therapy with one of the NOACs. Patients who stopped or didn't start NOAC treatment were asked about the reasons for non-adherence to anticoagulants use during visit 1 (6 months) and at PC (1 year).
Time Frame: Total - 1 year (two timepoints - 6 months (V1) and 1 year (PC))
Measure: Count of Participants; unit: Participants
Arm/Group | ANTEY
Number analyzed (Participants) | 7
Participants
  bleeding | 5
  cancellation by another doctor | 1
  high cost | 1

7. Secondary Outcome: Reasons for Stopping Oral Anticoagulants (Data From the Phone Contact)
Description: The study consisted of two visits half a year apart (V0, V1) and a phone contact (PC) one year after V0. During V0 all patients were recommended to start therapy with one of the NOACs. Patients who stopped NOAC treatmet were asked about the reasons for stopping oral anticoagulants (NOAC and warfarin) use during the phone contact.
Time Frame: Total - 1 year (two timepoints - 6 months (V1) and 1 year (PC)
Measure: Count of Participants; unit: Participants
Arm/Group | ANTEY
Number analyzed (Participants) | 18
Participants
  bleeding | 7
  cancellation by another doctor | 6
  high cost | 2
  others | 3

ADVERSE EVENTS:
Time Frame: 1 year
Description: All cause mortality - 4: 2 patients died of chronic diseases (heart failure, cancer), 1 patient had sudden cardiac death, and 1 patietnt died in an accident.
Arm/Group | ANTEY
All-Cause Mortality (participants affected / at risk) | 4/201
Serious Adverse Events (participants affected / at risk) | 21/201
Other Adverse Events (participants affected / at risk) | 30/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ANTEY (N=201)
Acute myiocardial infarction (Cardiac disorders) | 1 (1) — Non-fatal AMI
Unstable angina pectoris (Cardiac disorders) | 5 (5)
CHF decompensation (Cardiac disorders) | 5 (5) — Hospitalization due to CHF decompensation
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Paroxysm of atrial fibrillation (Cardiac disorders) | 5 (5) — Paroxysm of atrial fibrillation, emergency hospitalization
Stroke (Nervous system disorders) | 2 (2)
Bleeding in the retina (Eye disorders) | 1 (1) — Bleeding in the retina, emergency hospitalization
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) — Severe iron deficiency anaemia, emergency hospitalization
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ANTEY (N=201)
Bleeding (General disorders) | 18 (19) — Bleeding of different localization due to NOAC therapy, non-severe
Nausea (Gastrointestinal disorders) | 4 (4)
Urticaria (Immune system disorders) | 2 (2)
Obstipation (Gastrointestinal disorders) | 2 (2)
Hypothyroidism (Endocrine disorders) | 1 (1) — amiodarone-induced hypothyroidism
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Gynecomastia (Reproductive system and breast disorders) | 1 (1) — Spironolactone-induced gynecomastia
Arterial hypotension (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-12): https://cdn.clinicaltrials.gov/large-docs/17/NCT03790917/Prot_SAP_000.pdf